CLINICAL TRIAL: NCT03210246
Title: A Randomized, Double-blind, Parallel-group, Multi-center Study to Investigate the Pharmacodynamics and Pharmacokinetics of a Combined Oral Contraceptive Containing Levonorgestrel (LNG) and Ethinylestradiol (EE) When Given Together With Vilaprisan Over 3 Months in Healthy Women of Reproductive Age
Brief Title: Drug-drug Interaction Study: Influence of Vilaprisan on Pharmacodynamics (PD) and Pharmacokinetics (PK) of a Combined Oral Contraceptive (COC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 17670; 2016-004532-38 (EudraCT Number)
Record Dates: First submitted 2017-07-05; First posted 2017-07-06 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Clinical Trial ,Phase I
MeSH Terms: interventions — vilaprisan; ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COC + Vilaprisan (Experimental): COC + Vilaprisan (BAY 1002670)
  Interventions: Drug: Vilaprisan (BAY 1002670); Drug: Microgynon; Drug: Microgynon Placebo
- COC + Placebo (Placebo Comparator): COC + Placebo
  Interventions: Drug: Vilaprisan Placebo; Drug: Microgynon; Drug: Microgynon Placebo

INTERVENTIONS:
Drug: Vilaprisan (BAY 1002670) — Multiple doses of Vilaprisan for 3 cycles of 28 days each and 7 additional doses on the 7 days after cycle 3.
  Arms: COC + Vilaprisan
Drug: Vilaprisan Placebo — Multiple doses of placebo for 3 cycles of 28 days each and 7 additional doses on the 7 days after cycle 3.
  Arms: COC + Placebo
Drug: Microgynon — Multiple doses of Microgynon for 3 cycles of 21 days each (day 1-21)
Drug: Microgynon Placebo — For the treatment cycle 1-3, 7 doses of Microgynon placebo on Day 22-28 per cycle and after 3 treatment cycles 7 additional doses of Microgynon placebo on the 7 days after cycle 3 (day 84 - 91).

SUMMARY:
This study will be performed as a multi-center, randomized, double-blind study in 60 healthy women (2 groups of 30 women) to investigate ovarian activity during simultaneous intake of a COC (containing the estrogen EE and the progestin LNG) and the progesterone receptor modulator (PRM) vilaprisan.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female premenopausal subjects
* Age: 18 to 35 years (inclusive)
* Body mass index (BMI) : ≥18 and ≤30 kg/m²
* Non-smoker for 3 months (former smokers who quit smoking >3 months before the first study drug administration may be included)

Exclusion Criteria:

* Incomplete recovery from pre-existing disease for which it can be assumed that the absorption, distribution, excretion, and effect of the study drugs will not be normal
* presence or history of thrombophlebitis, venous or arterial thrombotic/thromboembolic events (e.g. deep venous thrombosis, pulmonary embolism, myocardial infarction) or of a cerebrovascular accident

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Number of subjects with ovulation (i.e. Hoogland score = 6) or risk of ovulation (Hoogland score = 5) | treatment day 57 to day 84
Number of subjects with a Hoogland score = 4 | treatment day 57 to day 84

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Germany (2):
  - Dinox GmbH Berlin, Berlin
  - CRS Clinical Research Services Berlin GmbH, Berlin